CLINICAL TRIAL: NCT03706443
Title: Tear Lipid Layer Thickness Changes With Use of Emollient and Non-Emollient Eye Drops
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Principal Investigator, Jennifer Fogt, Associate Professor, Ohio State University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2018H0433
Record Dates: First submitted 2018-10-11; First posted 2018-10-16 (Actual); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Dry Eye Syndromes; Keratoconjunctivitis Sicca; Lacrimal Apparatus Diseases; Keratoconjunctivitis; Eye Diseases; Keratitis; Corneal Disease; Ophthalmic Solution
MeSH Terms: conditions — Dry Eye Syndromes; Keratoconjunctivitis Sicca; Lacrimal Apparatus Diseases; Keratoconjunctivitis; Eye Diseases; Keratitis; Corneal Diseases

STUDY DESIGN:
Intervention Model Description: Single masked; randomized
Who Masked: Participant
Masking Description: Investigator instills known eye drop; masked to participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Systane® Complete (Active Comparator): All subjects are randomly assigned to arm one or arm two. Subjects are assigned to be treated with one drop of Systane® Complete, and the tear lipid layer thickness is to be measured at 15 minutes, 1, 2, 4, and 6 hours after instillation of the eye drop. Following a minimum of a 2-day washout, the same subjects will proceed to the second arm.
  Interventions: Other: Systane Complete
- Systane® Ultra (Active Comparator): All subjects are randomly assigned to arm one or arm two. Subjects are assigned to be treated with one drop of Systane® Ultra, and the tear lipid layer thickness is to be measured at 15 minutes, 1, 2, 4, and 6 hours after instillation of the eye drop. Following a minimum of a 2-day washout, the same subjects will proceed to the second arm.
  Interventions: Other: Systane Ultra

INTERVENTIONS:
Other: Systane Complete — Lubricant eye drop which is based on propylene glycol 0.6%. Used for temporary relief of burning and irritation due to dryness of the eye.
  Arms: Systane® Complete
Other: Systane Ultra — Lubricant eye drop which is based on polyethylene glycol 400 0.4% and propylene glycol 0.3%. Used for temporary relief of burning and irritation due to dryness of the eye.
  Arms: Systane® Ultra

SUMMARY:
Cross-over comparison of lipid layer thickness and dry eye symptoms with two artificial tear formulations.

DETAILED DESCRIPTION:
This study will objectively evaluate two US lubricant eye drop formulations produced by Alcon, INC. Systane® Ultra, a non-emollient eye drop, will be compared to Systane® Complete, an emollient eye drop, in subjects with dry eye symptoms and lipid layer thickness < 75 nm at baseline in a randomized, cross-over (masked subject) design. We seek to objectively evaluate the increase in lipid layer thickness from baseline at 15 minutes and 1, 2, 4 and 6 hours after each eye drop has been instilled. Non-invasive measurements of tear break-up time will be also conducted at each visit. Subjects will then be dispensed the emollient eye drop (Systane® Complete) for use four times daily for one month and return to the study site for final measurements of dry eye symptoms, lipid layer thickness, and tear break-up time. The Stroboscopic Video Color Microscope of King-Smith is used for non-invasive lipid layer thickness measurement, and the Oculus Keratograph (K5M) is used for non-invasive measurements of tear break-up time.

ELIGIBILITY:
Inclusion Criteria:

* Age - at least 30 years
* Good general health (defined by medication use that has not changed within the last month and the absence of medical conditions or treatments that are deemed confounding to the data as determined by the PI)
* Ability to give informed consent
* Willing to spend time for the study; approximately one hour for a screening visit and two eye drop exposure visits lasting approximately 6 hours each. Part 2 of the study will include using an eye drop of Systane® Complete 4x/day for 1 month and returning for one visit lasting approximately 1 hour.
* Either gender
* Any racial or ethnic origin
* SVCM tear lipid thickness ≤ 75 nm
* Contact lens wearers must refrain from lens wear for two days before the screening visit, including the day of the baseline visit, and during the entire study.

Exclusion Criteria:

* Use of any ocular prescription medication (such as but not limited to, glaucoma medications, anti-inflammatory eye drops and Restasis) used within 14 days of the screening visit or started prior to the measurement visit(s).
* Currently having punctal plugs inserted in lacrimal puncta
* Current eye disease, infection or inflammation that affects the surface of the eye such as, but not limited to moderate or greater blepharitis and ocular allergy. Clinically significant (active treatment) of blepharitis, Sjogren's disease or other systemic disease that could influence MGD, corneal, conjunctival, or eyelid abnormalities that could influence lipid layer thickness, conjunctivitis of any cause, ocular infection or systemic medication such as diuretics, SSRIs, that could influence tear secretion, or sensitivity to any of the ingredient in the eye drop being tested,
* Past eye surgery, such as, but not limited to, refractive surgery. Subjects who have had cataract removal surgery more than one year ago may be considered as potential subjects.
* Female subjects may not be pregnant or lactating. (Subject will be asked to self report these conditions.)
* Infectious diseases (for example, hepatitis, tuberculosis) or an immuno-suppressive disease (for example, HIV). (Subjects will be asked to self-report these conditions.)
* Inability to complete the screening and examination
* Inability to provide analyzable data. For example, subjects who cannot keep their eye open during the entire measurement interval (due to early blinking) or provide a readable eye image (due to eyelid laxity) or cannot sit still for 1 minute.

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-12-05 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Tear Lipid Layer Thickness | 1 minute
  Interference microscopy

SECONDARY OUTCOMES:
Tear Break-Up Time | 1 minute
  Oculus Keratograph (K5M)

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University College of Optometry, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No